CLINICAL TRIAL: NCT07201480
Title: Death Anxiety: Implications for Depression and Anxiety - An Experimental Study
Brief Title: Death Anxiety, Depression and Anxiety: An Experimental Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Roxana Cardos, PhD, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 430/ 30.04.2024
Record Dates: First submitted 2025-06-12; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Death Anxiety; Depression; Anxiety
Keywords: death anxiety; depression; anxiety; transdiagnostic
MeSH Terms: conditions — Necrophobia; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mortality Primed (Experimental): Participants in this arm will be instructed to answer two questions that are meant to bring to awareness thoughts about their mortality: "Please briefly describe the emotions that the thought of your death arouses in you." and "Jot down, as specifically as you can, what you think will happen to you physically as you die and once you are physically dead."
  Interventions: Behavioral: Mortality Salience Prompts
- Dental Pain Primed (Placebo Comparator): Participants in this arm will be instructed to answer two questions that may bring to mind thoughts and memories of dental pain: "Please briefly describe the emotions that the thought of dental pain arouses in you." and "Jot down, as specifically as you can, what you think happens to you physically as you experience dental pain and once you have physically experienced dental pain."
  Interventions: Behavioral: Dental Pain Prompts

INTERVENTIONS:
Behavioral: Mortality Salience Prompts — This intervention implies giving two prompts to participants, in a written format, while asking them to write out answers to the given prompts. The first prompt is: "Please briefly describe the emotions that the thought of your death arouses in you." The second prompt is "Jot down, as specifically as you can, what you think will happen to you physically as you die and once you are physically dead."
  Arms: Mortality Primed
Behavioral: Dental Pain Prompts — This intervention implies giving two prompts to participants, and requesting that participants write out their answers to these prompts. The first prompt is: "Please briefly describe the emotions that the thought of dental pain arouses in you." The second prompt is: "Jot down, as specifically as you can, what you think happens to you physically as you experience dental pain and once you have physically experienced dental pain."
  Arms: Dental Pain Primed

SUMMARY:
The goal of this experimental study is to investigate the transdiagnostic role of death anxiety in depression and anxiety symptoms in participants from the general population.

The main questions it aims to answer are:

1. Does the mortality salience task induce death anxiety?
2. Does the experimental group present an increase in depression and anxiety symptoms following the mortality salience task?

The investigators will compare the experimental condition to a control condition to see if the death anxiety induction is responsible for the expected increase in depression and anxiety symptoms.

The mortality salience prompt will be asking participants to elaborate on their thoughts and feelings surrounding death and dying, including what they think happens during death. The dental pain prompt will ask participants to do the same, only in regards to the thought of having dental pain.

Experimental group: participants will undergo a pen-and-paper writing task where they will be asked to answer two questions:

1. "Please briefly describe the emotions that the thought of your own death arouses in you."
2. "Jot down, as specifically as you can, what you think will happen to you physically as you die and once you are physically dead."

Control group:

1. "Please briefly describe the emotions that the thought of dental pain arouses in you."
2. "Jot down, as specifically as you can, what you think happens to you physically as you experience dental pain and once you have physically experienced dental pain."

DETAILED DESCRIPTION:
The purpose of this study is to investigate the role of death anxiety as a transdiagnostic factor in psychopathology. In this particular study, the investigators will examine whether increases in death anxiety - brought about by increasing the salience of death by use of a mortality salience prime lead to increases in levels of depression and anxiety.

Participants will provide their informed consent and will proceed to complete the measures of the study (pretest). Eligible participants will be randomly allocated to either the mortality salience group (experimental group), or the dental pain group (the control group). Participants will be blind to group allocation.

Two weeks after completing the pretest measures, the participants will come to the lab and undergo the experimental tasks, depending on the condition that they have been allocated to.

Experimental group: participants will undergo a pen-and-paper writing task where they will be asked to answer two questions

1. Please briefly describe the emotions that the thought of your own death arouses in you.
2. Jot down, as specifically as you can, what you think will happen to you physically as you die and once you are physically dead.

Control group: participants will undergo a pen-and-paper writing task where they will be asked to answer two questions

1. Please briefly describe the emotions that the thought of dental pain arouses in you.
2. Jot down, as specifically as you can, what you think happens to you physically as you experience dental pain and once you have physically experienced dental pain.

After the prime, participants will complete a distractor task, during which they will be asked to read a short, emotionally neutral text - a bogus scientific article, estimated to be a 5 minute read - and answer questions based on this text. Participants will be told that this task is done in order to assess text comprehension abilities. After completing the distractor task, participants will complete the study measures the second time (posttest).

Upon study completion, all participants will be debriefed in the lab, and the real purpose of the study will be explained to them.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Living in Cluj-Napoca (or otherwise willing and able to participate in the lab task)

Exclusion Criteria:

* Personality disorder diagnosis
* Psychotic disorder diagnosis
* Suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Collet-Lester Fear of Death Scale - Revised (CLFD-R) | Baseline (Day 1), After the experimental task (Day 14)
  The Revised version of the Collet-Lester Fear of Death Scale (CLFD-R) is a validated self-report instrument assessing fear and anxiety in regards to death and dying. The scale is comprised of 32 items that are answered from 1 (not at all) to 5 (very much) Possible scores range from 32 to 160. Higher scores indicate worse death anxiety.

SECONDARY OUTCOMES:
The Generalized Anxiety Disorder - 7 | Baseline (Day 1), After the experimental task (Day 14)
  The Generalized Anxiety Disorder 7-item Scale (GAD-7) is a validated self-report instrument that measures symptoms of generalized anxiety. It consists of 7 items rated on a 4-point scale from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 21. Higher scores indicate worse anxiety symptoms.
Patient Health Questionnaire - 9 | Baseline (Day 1), After the experimental task (Day 14)
  The Patient Health Questionnaire-9 (PHQ-9) is a validated self-report instrument assessing symptoms of depression. It consists of 9 items, each rated on a 4-point scale ranging from 0 (not at all) to 3 (almost every day). Total scores range from 0 to 27. Higher scores indicate worse depression symptoms.
State and Trait Anxiety Inventory - State subscale | Baseline (Day 1), After the experimental task (Day 14)
  The State-Trait Anxiety Inventory (STAI) is a validated self-report instrument assessing both state and trait anxiety. In this case, the State Anxiety subscale will be used, which is comprised of 20 items, each rated on a 4-point scale ranging from 1 (not at all) to 4 (very much so). Possible scores range from 20 to 80. Higher score indicate higher state anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
Will share IPD used in the results of the publication, upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD may be shared after publication upon request, with no end date.